CLINICAL TRIAL: NCT01307852
Title: Pilot Study to Evaluate In Vivo Plastic Scintillation Detectors for Real-Time Radiation Dosimetry During Prostate Cancer Radiotherapy
Brief Title: In Vivo Dosimetry During Prostate Cancer Radiotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0427; NCI-2011-00863 (Registry Identifier: NCI CTRP); 1R01CA120198-01A2 (NIH)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Disease
Keywords: Fiber optic radiation detectors; Enhanced endorectal balloon; Radiation treatment; Radiotherapy; External beam radiation; Dosimetry
MeSH Terms: conditions — Prostatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- In Vivo Dosimetry (Experimental): Modified endorectal device capable of real-time dose measurement during prostate radiation therapy
  Interventions: Device: Plastic Scintillation Detectors

INTERVENTIONS:
Device: Plastic Scintillation Detectors — Radiation detectors attached to rectal balloon for each CT scan done during each radiation treatment. Treatment delivery Monday through Friday for 7 weeks.

SUMMARY:
The goal of this clinical research study is to learn if a rectal balloon with attached radiation detectors can be used to help researchers monitor the dose of external beam radiation that is delivered to the prostate during treatment. This may help researchers better understand the side effects of radiation therapy, such as rectal bleeding, and may lead to changes in treatment planning or treatment delivery.

DETAILED DESCRIPTION:
As a part of your standard of care, you will have external beam radiation therapy. You will have a computerized tomography (CT) scan of the pelvis before the external beam radiation therapy.

For the CT scan, you will be given an enema to empty your bowel, and you will drink about 16 to 24 ounces of water to fill your bladder

A rectal balloon will then be inserted into your rectum and filled with either air or water. You will then have the CT scan. The CT scan should take about 45 minutes.

If you agree to take part in this study, very thin (millimeter-sized) radiation detectors will be attached to the rectal balloon during each of two CT scans per week you will have while you are receiving radiation. You may have additional CT scans (without the detector) each week if your doctor thinks it is needed.

The doses read by the radiation detectors will be compared to the doses that you were originally scheduled to receive after each radiation treatment and at the end of the study.

You will be off study after your final radiation treatment using the rectal balloon.

This is an investigational study. Up to 15 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients with prostate cancer who are undergoing routine radiation therapy for their prostate cancer, including post-prostatectomy patients.
2. The selection criteria will be limited to the patient's ability to withstand insertion of a rectal balloon and his willingness to participate in the study.
3. We will choose patients undergoing photon and proton treatments.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Measurement of True In Vivo Radiation to Rectal Wall During Prostate Radiotherapy | Twice a week for 7 week treatment.
  Twice a week in vivo measurements of radiation dose absorbed by the rectal wall during intensity-modulated radiotherapy (IMRT) of prostate.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Beddar, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org